CLINICAL TRIAL: NCT01850550
Title: Impact of Volunteer Peer-Led Intervention for Weight Control in Primary Care
Acronym: KL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Kraschnewski, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KL2; UL1TR000127 (NIH); KL2TR000126 (NIH)
Record Dates: First submitted 2013-04-29; First posted 2013-05-09 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Weight Loss
Keywords: Weight loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants in the control condition will be given written information at the baseline visit from the NIH website "Aim for a Healthy Weight" to provide a basic understanding of weight loss and access to basic online resources, but will not participate in group weight loss sessions with peer leaders.
- Weight Loss Groups (Experimental): Participants in this arm will receive peer-led facilitation within groups using an adaptation of the Diabetes Prevention Program.
  Interventions: Behavioral: Weight loss Groups

INTERVENTIONS:
Behavioral: Weight loss Groups — The intervention will consist of 12 weekly one-hour weight loss sessions led by successful volunteer peers. Participants are provided with a modified version of the Diabetes Prevention Program manual and are mentored by peer leaders at weight loss sessions.
  Arms: Weight Loss Groups

SUMMARY:
The specific objective of this research proposal is to determine the short-term efficacy of a primary care-based weight control intervention in which successful volunteer peers deliver a group-based program.

The purpose of the study is to conduct a pilot randomized controlled trial (RCT) of a successful volunteer peer-led weight control program compared to a control condition to determine intervention efficacy at 3 months. Six peer leaders from 2 primary care clinics will be recruited and trained to conduct the intervention. Overweight and obese patients (n=80) will be recruited (randomized by individual) to determine weight loss at 3 months (primary outcome). The program consists of 12 weekly weight loss sessions led by a successful volunteer peer leader using an adaptation of the Diabetes Prevention Program to help participants lose weight.

DETAILED DESCRIPTION:
The intervention will consist of 12 weekly one-hour weight loss sessions led by successful volunteer peers. The initial weight loss session will be conducted by the peer leaders with oversight by the PI. This session will serve to introduce the program and give an overview of program. The remaining sessions, conducted by co-peer leaders, will utilize an adaptation of the Diabetes Prevention Program. This adaptation allows for use in a group setting and facilitation by a lay individual.

Control Condition: Participants in the control condition will be given written information at the baseline visit from the NIH website "Aim for a Healthy Weight" to provide a basic understanding of weight loss and access to basic online resources. We expect that use of the website may result in some weight loss. However, similar information-only interventions have had a very small effect, which is accounted for in the sample size calculation.

ELIGIBILITY:
PEER Inclusion Criteria:

* Successful at volitional weight loss, defined as at least 10% of their initial body weight and maintenance for ≥ 1 year
* Fluently speak and read English
* Willing to volunteer 1 hour each week as a group leader
* Able and willing to give informed consent.
* Must have internet access

Participant Inclusion Criteria:

* Fluently speak and read English
* Able and willing to give informed consent
* Body Mass Index > 25 and < 45
* Interested in participating in weekly group sessions for weight loss
* Must have internet access

Exclusion Criteria:

* Current or planned pregnancy within the next year
* Medical or other contraindications to weight loss, including, but not limited to, history of:

  1. Myocardial infarction
  2. Stroke
  3. Unstable angina
  4. Congestive heart failure
  5. Cancer (except non-melanoma skin cancer)
* History of gastric bypass surgery or scheduled surgery for this purpose
* Current use of prescription medication for weight loss
* Weight loss of > 5% of current body weight in previous 6 months
* Contraindications to weight loss
* Evidence of severe cognitive impairment or major psychiatric illness
* Plans to move in the next 6 months
* Answering yes to any question on the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Kraschnewski, MD, MPH, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Weight Loss Groups
Started | 40 | 40
Completed | 40 | 37
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Weight Loss Groups | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Weight
Description: We will assess our participants to evaluate the percent change in weight over the 12 week period of the study using a scale.
Time Frame: 12 weeks after initial consent
Measure: Mean (Full Range); unit: percent weight change
Arm/Group | Control | Weight Loss Groups
Number analyzed (Participants) | 40 | 37
percent weight change | -1.27 [-16.8 to 3.99] | -2.76 [-10.37 to 4.01]

2. Secondary Outcome: BMI
Description: Change in BMI from baseline to follow up will be assessed using a scale and stadiometer.
Time Frame: 12 weeks after initial consent
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Control | Weight Loss Groups
Number analyzed (Participants) | 40 | 37
kg/m^2 | -0.04 [-3.02 to 1.50] | -0.11 [-4.03 to 1.33]

3. Secondary Outcome: Blood Pressure
Description: Blood pressure will be recorded using an OMRON automatic blood pressure cuff.
Time Frame: 12 weeks after initial consent
Reporting Status: Not Posted

4. Secondary Outcome: Physical Activity
Description: Assessed by the International Physical Activity Questionnaire
Time Frame: 12 weeks after initial consent
Reporting Status: Not Posted

5. Secondary Outcome: Dietary Intake
Description: Assessed using the NCI Dietary History Questionnaire
Time Frame: 12 weeks after initial consent
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Weight Loss Groups
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
This was a pilot study. No other limitations noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes